CLINICAL TRIAL: NCT05050643
Title: Improving Care for Complex, High-Risk Patients in Primary Care (QUE 20-018)
Brief Title: High-Risk Veteran Initiative
Acronym: RIVET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Veterans Health Administration Office of Primary Care (Unknown); Veterans Health Administration Office of Patient Centered Care & Cultural Transformation (Unknown); US Department of Veterans Affairs (U.S. Federal Agency); Veterans Integrated Service Network 10 (Unknown); Veterans Integrated Service Network 12 (Unknown); VA MidSouth Healthcare Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 21-005
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Multimorbidity
Keywords: Primary Health Care; Multimorbidity; Medication Adherence; Needs Assessment; Mentoring
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a mixed-methods type 3 hybrid implementation-effectiveness evaluation using a Concurrent Stepped Wedge design to compare two implementation strategies to increase adoption of the EBPs in primary care in 16 sites: Evidence-Based Quality Improvement (EBQI)-Individual Consultation (EBQI-IC) and EBQI-Learning Collaborative (EBQI-LC). Each VISN will implement a single EBP [Comprehensive Assessment and Care Planning (CACP) for High-Risk Veterans or Phone-Based Health Coaching for Medication Adherence (HCMA)]. Implementation strategies will be randomized by site. Time periods without active implementation will serve as the usual care periods for both EBQI conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CACP-EBQI-IC (Active Comparator): Individual (ongoing) consultation (IC), often described as coaching or supervision, is endorsed by implementation experts as an effective implementation strategy for EBP #1, Comprehensive Assessment and Care Planning (CACP) for High-Risk Veterans.
  Interventions: Other: EBQI-IC
- CACP-EBQI-LC (Active Comparator): Learning collaboratives (LC) are widely used in healthcare settings, as an effective implementation strategy. The LC will be used to increase uptake of EBP #1, Comprehensive Assessment and Care Planning (CACP) for High-Risk Veterans.
  Interventions: Other: EBQI-LC
- HCMA-EBQI-IC (Active Comparator): Individual (ongoing) consultation (IC), often described as coaching or supervision, is endorsed by implementation experts as an effective implementation strategy for EBP # 2,Phone-Based Health Coaching for Medication Adherence (HCMA).
  Interventions: Other: EBQI-IC
- HCMA-EBQI-LC (Active Comparator): Learning collaboratives (LC) are widely used in healthcare settings, as an effective implementation strategy. The LC will be used to increase uptake of EBP # 2,Phone-Based Health Coaching for Medication Adherence (HCMA).
  Interventions: Other: EBQI-LC

INTERVENTIONS:
Other: EBQI-IC — Individual (ongoing) consultation (IC), often described as coaching or supervision, is endorsed by implementation experts as an effective implementation strategy
  Other Names: Individual Consultation
  Arms: CACP-EBQI-IC; HCMA-EBQI-IC
Other: EBQI-LC — A Learning Collaborative is a systematic approach to process improvement based on the Institute for Healthcare Improvement Breakthrough Series Collaborative model. During the Collaborative, organizations will test and implement system changes and measure their impact. They will share their experiences to accelerate learning and broader implementation of best practices.
  Other Names: Learning Collaborative
  Arms: CACP-EBQI-LC; HCMA-EBQI-LC

SUMMARY:
Veterans at high-risk for hospitalization, including those with complex care needs, represent a large population of VHA patients who often do not receive evidence-based primary care practices that would help them avoid the hospital and improve their health. The high-RIsk VETerans (RIVET) Program will implement evidence-based practices that can support VHA Primary Care teams to deliver more comprehensive and patient-centered care, better strategies to manage medications, and avoid unnecessary hospitalizations. The RIVET Program is designed to find the most effective approaches to increasing use of evidence-based practices for high-risk Veterans in primary care, provide rapid data feedback to VHA on high-risk patient care, build capacity for the implementation of evidence-based practices, and train future leaders in high-risk Veteran care.

DETAILED DESCRIPTION:
The top 5% of Veterans at the highest risk for hospitalizations account for almost 50% of VHA healthcare costs, have significant multimorbidity, and are also at high risk for poor health outcomes. In the VHA, most (88%) high-risk patients are managed by general primary care teams (i.e., Patient-Aligned Care Teams; PACTs). Few PACTs, however, have implemented evidence-based practices (EBPs) known to address the most common issues among high-risk Veterans. Some evidence indicates that usual implementation strategies, such as dissemination of toolkits and training are not effective for improving uptake of EBPs. The most effective implementation strategies to achieve evidence-based care for high-risk patients, however, are unknown.

The overall impact goal of the high-RIsk VETerans (RIVET) QUERI Program is to improve VHA primary care capacity to provide comprehensive, evidence-based care for complex, high-risk Veterans. The investigators will test 2 implementation strategies to evaluate their impact on the uptake of two separate EBPs. These EPBs are 1) Comprehensive Assessment and Care Planning (CACP), and 2) Phone-Based Health Coaching for Medication Adherence (HCMA). CACP is based on the Comprehensive Geriatric Assessment and guides teams in systematically addressing patients' cognitive, functional, and social needs through a comprehensive care plan. HCMA addresses common challenges to medication adherence using a patient-centered approach through virtual encounters. Both comprehensive assessments and health coaching have demonstrated efficacy in randomized, controlled trials and have been implemented by two of the national partners in geriatrics and Whole Health teams. However, both EBPs have had low uptake in primary care. Implementing these practices in primary care has the potential to improve quality of care for the large majority of high-risk Veterans. The investigators will conduct a mixed methods type 3 hybrid effectiveness-implementation design to test the effectiveness of EBQI-IC and EBQI-LC versus usual care (national tool dissemination and training efforts) in at least 16 sites in multiple VISNs using a Concurrent Stepped Wedge design (Aim 2). The primary outcome is proportion of eligible high-risk patients that receive each EBP. The investigators will use the Practical, Robust Implementation and Sustainability Model (PRISM) framework to compare and evaluate Reach, Effectiveness, Adoption, Implementation, and costs. The investigators will then assess the Maintenance/sustainment and spread of both EBPs in primary care across all sites after the active 18-month implementation period (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

Any VA site nationwide

Exclusion Criteria:

Not a VA site nationwide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the proportion of team-assigned primary care patients in the upper 90th percentile of acute hospitalization risk (identified via VA CAN score) who received the Evidence Based Practice (EBP) | 18
  This primary outcome aims to measure reach of the evidence practices to implement the EBP.

SECONDARY OUTCOMES:
Number of PACT encounters from social worker, pharmacist, nurse and integrated mental health | 18 months
  This secondary outcome will measure the impact of EBPs on the proximal care process.
Number of encounters from PACT pharmacist, social worker, nurse and integrated mental health | 18 months
  This secondary outcome will measure the impact of EBPs on the proximal care process.
Comprehensiveness of Care questions from the RIVET Patient Survey- consisting of three items, which was sourced from the SHEP | 18 months
  This secondary outcome will measure patient impact due to EBPs.
Self-Management Support questions from the RIVET Patient Survey- sourced from the SHEP, which is two items in the survey. | 18 months
  This secondary outcome will measure patient impacts due to EBPs .
PACT provider perceived support for high-risk patient care questions from the RIVET Clinician Survey- three survey items assessing confidences, skills and strain/satisfaction with caring for high-risk patients | 18 months
  This secondary outcome will measure patient impacts of EBP#1 (CACP).
Providers Discuss Medication Decisions (Patient Survey) | 18 months
  This secondary outcome will measure patient impacts of due to EBPs.
Self-Management Support (Patient Survey) | 18 months
  This secondary outcome will measure patient impacts of due to EBPs.
Total number of ambulatory care-sensitive and acute hospitalizations | 18 months
  This secondary outcome will measure clinical quality due to EBPs.
Total number of ambulatory care-sensitive and and emergency department visits | 18 months
  This secondary outcome will measure clinical quality due to EBPs.
Patient self-reported medication adherence This survey is a 3-item scale developed and validated in Veteran populations | At the beginning and end of 18-month implementation period
  This survey is a 3-item scale developed and validated in Veteran populations.
Adherence to chronic medications (diabetes, hypertension, hyperlipidemia, mental health) (VA Pharmacy Data) | The 18-month implementation period
  This secondary outcome will measure clinical quality outcome of EBP#2(HCMA). Medications will be calculated via VA pharmacy fill data using Proportion of Days Covered (PDC).
Adoption of Evidence Based Practice (EBP) | 30-months
  Proportion of staff trained on EBPs.
HEDIS measures for diabetes, hypertension, hyperlipidemia management | The 18-month implementation period
  This secondary outcome will measure clinical quality outcome due to EBPs.
Fidelity | 18 months
  The fidelity assessment tool draws from data collected from key stakeholder interviews , implementation facilitation logs , administrative documents, and weekly time diaries. The team will apply criteria to rate sites as high-, medium-, or low-fidelity on the EBQI elements.
EBP Fidelity | 18 months
  A composite EBP fidelity measure for each EBP will be assessed by percent of items completed.
Implementation costs | 18 months
  Implementation Core staff time spent in various implementation activities
Facility adopting cost | 18 months
  Cost calculated from time incurred by facilities adopting the EBPs

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn T Chang, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA; Susan E Stockdale, PhD MA, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (3):
- United States (3):
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez EE, Rosland AM, Stockdale SE, Reddy A, Wong MS, Torrence N, Huynh A, Chang ET. Implementing evidence-based practices to improve primary care for high-risk patients: study protocol for the VA high-RIsk VETerans (RIVET) type III effectiveness-implementation trial. Implement Sci Commun. 2024 Jul 15;5(1):75. doi: 10.1186/s43058-024-00613-9. PMID 39010160